CLINICAL TRIAL: NCT02407262
Title: Potential Benefits of Black Seed Oil Supplementation on Asthma Inflammation and Outcomes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Abdulrahman Koshak, Postgraduate researcher, University College, London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6419/002
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Asthma
Keywords: asthma; black seed; Nigella sativa; supplementation
MeSH Terms: conditions — Asthma | interventions — Nigella sativa oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Active Comparator): Black seed oil capsules
  1g/day for 4 weeks
  Interventions: Dietary Supplement: Black seed oil
- Placebo (Placebo Comparator): Placebo (olive oil) capsules
  1g/day for 4 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Black seed oil
  Other Names: Nigella sativa oil
  Arms: Treatment
Other: Placebo — vegetable oil
  Arms: Placebo

SUMMARY:
Traditionally, Black Seed (Nigella sativa) is a well-known food supplement and herbal product that has a wide range of medical claims (including asthma) that originate from different historical backgrounds. Today in the era of Evidence-based medicine, it is hard to accept those traditional medical claims of medicinal plants without valid scientific experiments. Thus, randomized clinical trials is important to rational the uses of herbal products.

Asthma is a common chronic disorder of the airways, characterized by variable reversible and recurring symptoms related to airflow obstruction, bronchial hyper-responsiveness, and underlying inflammation. In Saudi Arabia, Asthma is considered one of the leading chronic diseases affecting more than 2 million Saudi citizens. The global Asthma Report 2014 considered Asthma as an epidemic disease probably affecting about 334 million people worldwide and becoming a global health priority.

This project investigates the use of herbal products to enhance asthma control in Saudi Arabia. In this context, Black Seed is one of the common herbal products used traditionally for asthma in the Saudi region. Black seed is a common unconventional therapy used among 10% of Asthmatic patients in King Abdulaziz Medical city, Riyadh. In fact, there are some pre-clinical evidence and preliminary clinical studies support the usefulness of Black seed in Asthma and its underlying causes

ELIGIBILITY:
Inclusion Criteria:

* Adult male/female (age 18-65 years),
* asthmatic patient with Asthma Control Test (ACT) score <25
* No severe asthma exacerbation in the last 4 weeks
* Able to obtain consent

Exclusion Criteria:

* Patients with serious co-morbid conditions such as; cancer, renal, hepatic, cardio-vascular, gastrointestinal diseases, mental health conditions and respiratory disorder such as TB and COPD.
* Smoking history
* Pregnant women
* Currently taking any form of Black seed.
* Known history of hypersensitivity to Black seed.
* Taking medications that may interact with black seed supplement: Anticoagulant/Antiplatelet, CNS depressants, and Immunosuppressant drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Asthma Control Test (ACT) | 4 weeks

SECONDARY OUTCOMES:
Serum inflammatory mediators | 4 weeks
  IL4, IL5, IL8, IL6, IL10, IL13, TNFa, IFN-g
Total IgE | 4 weeks
Complete blood count (CBC) | 4 weeks
  Mainly blood eosinophils
Pulmonary function test (predicted FEV1%) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Heinrich, PhD, Principal Investigator — University College, London
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

REFERENCES:
- [Background] Al Moamary MS. Unconventional therapy use among asthma patients in a tertiary care center in Riyadh, Saudi Arabia. Ann Thorac Med. 2008 Apr;3(2):48-51. doi: 10.4103/1817-1737.39636. PMID 19561905
- [Background] Al-Moamary MS, Alhaider SA, Al-Hajjaj MS, Al-Ghobain MO, Idrees MM, Zeitouni MO, Al-Harbi AS, Al Dabbagh MM, Al-Matar H, Alorainy HS. The Saudi initiative for asthma - 2012 update: Guidelines for the diagnosis and management of asthma in adults and children. Ann Thorac Med. 2012 Oct;7(4):175-204. doi: 10.4103/1817-1737.102166. PMID 23189095
- [Background] Boskabady MH, Javan H, Sajady M, Rakhshandeh H. The possible prophylactic effect of Nigella sativa seed extract in asthmatic patients. Fundam Clin Pharmacol. 2007 Oct;21(5):559-66. doi: 10.1111/j.1472-8206.2007.00509.x. PMID 17868210
- [Background] Salem ML. Immunomodulatory and therapeutic properties of the Nigella sativa L. seed. Int Immunopharmacol. 2005 Dec;5(13-14):1749-70. doi: 10.1016/j.intimp.2005.06.008. Epub 2005 Jul 1. PMID 16275613
- [Background] Lebling, R., & Pepperdine, D. (2006). Natural Remedies of Arabia (p. 223). Stacey Intl.
- [Background] Salama, R. (2010). Clinical and Therapeutic Trials of Nigella Sativa. TAF Preventive Medicine Bulletin, 9(5), 513-522.
- [Background] Singh BB, Khorsan R, Vinjamury SP, Der-Martirosian C, Kizhakkeveettil A, Anderson TM. Herbal treatments of asthma: a systematic review. J Asthma. 2007 Nov;44(9):685-98. doi: 10.1080/02770900701247202. PMID 17994396
- [Derived] Koshak A, Wei L, Koshak E, Wali S, Alamoudi O, Demerdash A, Qutub M, Pushparaj PN, Heinrich M. Nigella sativa Supplementation Improves Asthma Control and Biomarkers: A Randomized, Double-Blind, Placebo-Controlled Trial. Phytother Res. 2017 Mar;31(3):403-409. doi: 10.1002/ptr.5761. Epub 2017 Jan 17. PMID 28093815